CLINICAL TRIAL: NCT07324785
Title: The Role and Mechanism of SphK1/S1P/FOXO1 Axis Regulating KATP Channel Mediated Gastric Smooth Muscle Dysfunction in Diabetes Gastroparesis
Brief Title: Correlation Between Advanced Glycation End Products and Gastric Motility Disorder in Diabetes Gastroparesis
Status: Not yet recruiting | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025ky077
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Gastroparesis
Keywords: Diabetic gastroparesis; Advanced glycation end products

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — The gastric tissue, serum, and plasma will be retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic gastroparesis group: 1. Meet the diagnostic criteria for diabetes; 2. Presence of symptoms (see assessment of Gastroparesis Cardinal Symptom Index); 3. Age range from 18 to 75 years old; 4. Voluntarily participate and sign an informed consent form.
- control group: 1. No history of diabetes; 2. No symptoms (see assessment of Gastroparesis Cardinal Symptom Index); 3. Age range from 18 to 75 years old; 4. Voluntarily participate and sign an informed consent form.

SUMMARY:
This study is a prospective observational study. The study will explore the correlation between advanced glycation end products and gastric motility disorder in diabetic gastroparesis（DGP) through the collection of blood and gastric tissue samples and relevant data of patients with DGP and control group patients without diabetes history and gastroparesis symptoms.

DETAILED DESCRIPTION:
This study will collect the gastric smooth muscle tissue and serum of patients with diabetic gastroparesis（DGP) and control group patients without diabetes history and gastroparesis symptoms, and collect the following patient related information: age, gender, height, weight, fasting blood glucose, diabetes course, glycosylated hemoglobin, fasting C-peptide, serum creatinine, and electrogastrogram results.

The study will compare the score of gastroparesis cardinal symptom index scale and electrogastrogram results of patients with DGP and and control group patients without diabetes history and gastroparesis symptoms, detect and compare the difference in the expression of contractile protein in the muscle layer of gastric tissue of the two groups, detect and compare the difference in advanced glycation end products (AGEs) of serum and gastric tissue of the two groups, and analyze the correlation between serum and gastric tissue AGEs and clinical symptoms. Through the above results, we will clarify the correlation between AGEs and gastric motility disorders in DGP.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria for diabetes gastroparesis group: 1. Meet the diagnostic criteria for diabetes; 2. Presence of symptoms (see assessment of Gastroparesis Cardinal Symptom Index); 3. Age range from 18 to 75 years old; 4. Voluntarily participate and sign an informed consent form.

Inclusion Criteria for control group: 1. No history of diabetes; 2. No symptoms (see assessment of Gastroparesis Cardinal Symptom Index); 3. Age range from 18 to 75 years old; 4. Voluntarily participate and sign an informed consent form.

-

Exclusion Criteria: Exclusion Criteria for diabetes gastroparesis group and control group: 1. Currently taking prokinetic drugs, anticholinergic drugs, and dopamine drugs that may affect gastric motility; 2.Has a history of gastrointestinal surgery; 3. Pregnant or preparing to conceive; 4. There are neurological disorders such as Parkinson's disease that affect gastrointestinal function. 5. Outlet obstruction caused by organic lesions in the pylorus;

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic gastroparesis and control group patients in Northern Jiangsu People's Hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Gastroparesis Cardinal Symptom Index (GCSI) score | The day when the subjects were enrolled
  The Gastroparesis Cardinal Symptom Index (GCSI) is a patient-reported outcome measure used to assess the severity of gastroparesis symptoms. It consists of nine items grouped into three subscales: postprandial fullness/early satiety, nausea/vomiting, and bloating. Patients rate the severity of each symptom on a scale from 0 (no symptom) to 5 (very severe). The GCSI score is calculated as an average score of all three symptom categories. It is a reliable and valid tool for evaluating symptom severity and treatment effectiveness in clinical trials and other studies

SECONDARY OUTCOMES:
The results of electrogastrogram | On the day of the subject's electrogastrogram examination
  The results of electrogastrogram mainly include the frequency and amplitude of slow waves, the proportion of gastric electrical rhythm disturbances, and the proportion of normal slow waves in the electrogastrogram.

OTHER OUTCOMES:
Content of advanced glycation end products in serum and gastric tissue | After obtaining serum and gastric tissue
  Detection of advanced glycation end products in serum and gastric tissue by western blot and ELISA
Expression level of gastric tissue contractile protein | After obtaining serum and gastric tissue
  Detection of the expression of gastric tissue contractile protein by western blot and qRT-PCR
Heart rate variability | On the day of the subject's electrocardiogram signal recording
  Perform heart rate variability analysis on the recorded electrocardiogram signals.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhu, Doctor's degree, Principal Investigator — Northern Jiangsu People's Hospital
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The data underlying this article will not be shared as it contains patients' information and data.